CLINICAL TRIAL: NCT00565682
Title: Pain Post Abdominal Laparoscopy Prevention With Arcoxia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Vozandez (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Eduardo Noboa, Hospital Vozandez
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOLAAR
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Laparoscopic Surgery for Appendicitis; Laparoscopic Surgery for Cholecystitis; Laparoscopic Surgery for Ovarian Cysts
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Etoricoxib 120 mg
  Interventions: Drug: etoricoxib 120 mg

INTERVENTIONS:
Drug: etoricoxib 120 mg — etoricoxib 120 mg, tablet, orally, OD
  Other Names: Arcoxia

SUMMARY:
To test the analgesic efficacy of etoricoxib used before a surgical procedure compared to the already known effect when administered after such a procedure. Patient will be receiving either etoricoxib or the respective placebo one hour before surgery, then two hours after those receiving the active will receive placebo and those that received placebo will be given etoricoxib. Pain score measurements will be performed sequentially. Rescue medication will be available all the time.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary acceptance to participate in the study and signed the informed consent form
* Age older than 18 years old and younger than 70 years
* Diagnosis of appendicitis, cholecystitis or ovarian cysts suitable of laparoscopic surgery

Exclusion Criteria:

* Age less than 18 years or older than 70 years.
* Laparoscopic procedures for diagnostic purposes.
* Current use of anticoagulants.
* Known hypersensitivity to etoricoxib or its components.
* History of a CABG or MI (less than 1 year)
* History of unstable angina (over the past six months).
* Current inflammatory bowel disease.
* Uncontrolled hypertension or heart failure
* Renal dysfunction/impairment (creatinine clearance < 30ml/min)
* Cirrhosis or severe hepatic dysfunction
* Any degree of dehydration (mild to severe)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To measure the amount of rescue medication (opioid) needed to relief | Every hour after surgery

SECONDARY OUTCOMES:
To determine the overall analgesic effect using the visual analog scale (VAS) | Every hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Noboa, MD, Principal Investigator — Hospital Vozandez